CLINICAL TRIAL: NCT00267228
Title: Funen Anorexia Nervosa Study - Retrospective Cohort Study and 10 Year Follow-up Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Other Study IDs: 018
Record Dates: First submitted 2005-12-19; First posted 2005-12-20 (Estimated); Last update posted 2007-03-23 (Estimated); Status verified 2007-03

CONDITIONS: Anorexia Nervosa; Eating Disorder
Keywords: Anorexia Nervosa; Eating disorder; Quality of life
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study are:

1. Retrospectively to study the clinical characteristics and features (somatic, psychological and social variables) of patients treated in Center for Eating Disorders, Odense University Hospital 1994-2004.
2. To study the predictive power of the psychosocial and morphometric data with regard to drop outs, relapse and outcome.
3. To investigate eating habits, social functions and quality of life in weight recovered and chronicly ill patients with eating disorder.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated in Center for Eating Disorders, Odense University Hospital 1994 - 2004.

Exclusion Criteria:

* Patients, who according to the primary clinical evaluation was found not to suffer from eating disorder.
* Patients who at admission did not live in the Funen County.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2006-02

CONTACTS AND LOCATIONS:
Overall Officials: René K. Stovring, MD, PhD, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Frolich J, Winkler LA, Abrahamsen B, Bilenberg N, Hermann AP, Stoving RK. Assessment of fracture risk in women with eating disorders: The utility of dual-energy x-ray absorptiometry (DXA)-Clinical cohort study. Int J Eat Disord. 2020 Apr;53(4):595-605. doi: 10.1002/eat.23245. Epub 2020 Feb 12. PMID 32048754
- [Derived] Frolich J, Winkler LA, Abrahamsen B, Bilenberg N, Hermann AP, Stoving RK. Fractures in women with eating disorders-Incidence, predictive factors, and the impact of disease remission: Cohort study with background population controls. Int J Eat Disord. 2020 Jul;53(7):1080-1087. doi: 10.1002/eat.23223. Epub 2020 Jan 10. PMID 31922277